CLINICAL TRIAL: NCT03200548
Title: Acupressure for Persistent Fatigue in Systemic Lupus Erythematosus Patients
Brief Title: Acupressure for Fatigue in Systemic Lupus Erythematosus
Acronym: AcuSLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low participant recruitment and retention
Sponsor: Suzanna Zick (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Suzanna Zick, Co-Director of Integrative Family Medicine Research Associate Professor Department of Family Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00127631
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-06

CONDITIONS: Fatigue; Lupus Erythematosus, Systemic; Pain, Chronic; Quality of Life; Sleep
MeSH Terms: conditions — Fatigue; Lupus Erythematosus, Systemic; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The investigators propose to perform a randomized, single-blind parallel clinical trial. This will be parallel design with four arms (relaxing acupressure plus usual care, stimulating acupressure plus usual care, sham acupressure plus usual care and usual care alone) for persistent fatigue in SLE.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The three acupressure formulas will be labeled acupressure set "A", set "B", and set "C". Acupressure educators, outcome assessors, study participants, and study investigators (who will not interact with any of the study participants) will be blinded as to acupressure allocation. Only after data analysis is completed will the randomization code be unblinded. Those randomized to usual care will know that they are not receiving acupressure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Relaxing acupressure plus usual care (Experimental): There is a set of unilateral and bilateral acupoints that will be stimulated for 3 minutes per point giving a total treatment time of about 30 minutes daily.The "True Acupressure" points were chosen based on a TCM theory for treating insomnia.
  Interventions: Behavioral: Relaxing acupressure plus usual care
- Stimulating acupressure plus usual care (Experimental): There is a set of unilateral and bilateral acupoints that will be stimulated for 3 minutes per point giving a total treatment time of about 30 minutes daily. Acupoints were chosen by consensus of 4 acupressure practitioners and based on a previous study design in students with sleep disturbances as well as TCM theory for treating insomnia and fatigue.
  Interventions: Behavioral: Stimulating acupressure plus usual care
- Sham acupressure plus usual care (Sham Comparator): There is a set of unilateral and bilateral acupoints that will be stimulated for 3 minutes per point giving a total treatment time of about 30 minutes daily. None of these points are on meridians nor are they on actual points. They were chosen to be in the same general body quadrant as the true points.
  Interventions: Behavioral: Sham acupressure plus usual care
- Usual care (Placebo Comparator): Participants will be asked to continue following their healthcare providers' instruction for chronic SLE management. We anticipate that most women will be treated per the American College of Rheumatology clinical guidelines. Participants will be asked to continue any current treatment and not to start or stop treatments including acupuncture/acupressure over the course of the study. All treatments for pain will be recorded.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Relaxing acupressure plus usual care — Experimental group. Self-administered acupressure is one possible safe, self-management technique for which may be effective for improving fatigue as well as physical and psychosocial functioning in several chronic disease populations. Acupressure, a technique derived from acupuncture, is a component of Traditional Chinese Medicine (TCM) in which pressure is applied to specific acupoints on the body using a finger or small device, to treat disease.
  Arms: Relaxing acupressure plus usual care
Behavioral: Usual care — Negative control group. Participants are asked to carry on with their usual management practices and habits.
  Arms: Usual care
Behavioral: Stimulating acupressure plus usual care — Experimental group. Self-administered acupressure is one possible safe, self-management technique for which may be effective for improving fatigue as well as physical and psychosocial functioning in several chronic disease populations. Acupressure, a technique derived from acupuncture, is a component of Traditional Chinese Medicine (TCM) in which pressure is applied to specific acupoints on the body using a finger or small device, to treat disease.
  Arms: Stimulating acupressure plus usual care
Behavioral: Sham acupressure plus usual care — Positive control group. Chosen pressure points are not known to be effective.
  Arms: Sham acupressure plus usual care

SUMMARY:
Systemic lupus erythematosus (SLE) is a complex autoimmune disease characterized by involvement of multiple organs with a female to male ratio of 12:1 with the highest incidence reported in women of child bearing age (15-44 years). In general, advances in diagnosis and management have led to significant improvements in outcomes. However, fatigue remains a challenging and prevalent issue for SLE patients.

The investigators aim to determine the feasibility of recruiting and conducting acupressure in fatigued persons with lupus; to explore the effect of two distinct acupressure formulas (relaxing and stimulating) plus usual care versus sham acupressure plus usual care and usual care alone on severity and impact of chronic fatigue (as measured by the Brief Fatigue Inventory) as well as quality of life, sleep and pain.

DETAILED DESCRIPTION:
Self-administered acupressure is one possible safe, self-management technique that may be effective for improving fatigue as well as physical and psychosocial functioning in several chronic disease populations. Acupressure, a technique derived from acupuncture, is a component of Traditional Chinese Medicine (TCM) in which pressure is applied to specific acupoints on the body using a finger or small device, to treat disease. Our prior research demonstrated that acupressure, self-administered by women with breast cancer, significantly reduced clinically significant fatigue by approximately one-third in fatigued breast cancer survivors and was superior to standard therapies. Moreover these self-rated improvements were maintained up to one month after treatment was discontinued.

However, impact on other chronic disease populations with fatigue is unknown. To explore this intervention in SLE, the investigators are conducting a pilot randomized clinical trial among 72 SLE patients with established fatigue. The study will take place over the course of 12 weeks, including 5 participant interactions.

After completing the initial screening phone call, participant eligibility will be determined. If a participant is found ineligible then his or her participation in the study will end. If a participant is found eligible he or she may continue participation by attending the baseline visit during which participants will be randomized into one of four groups, three of which will be some type of acupressure and one which will be usual care.

In three of these groups participants will be taught how to perform acupressure and where your acupressure points are located by study staff members that have been trained by a certified acupressure practitioner. Each treatment group uses a different set of acupressure points and is instructed how to effectively stimulate those different points. The study staff member will demonstrate on the participant how much pressure to apply at an acupressure point and will observe the participant locating each acupressure point. Participants will also be given information to take home showing them where these acupressure points are placed on the body.

As part of this study, participants will be asked to attend 2 visits, answer phone calls or emails, and (if randomized to a treatment group) perform acupressure daily. There is also a follow-up visit or telephone call conducted at least 4 weeks after the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Report chronic (> 3 months) clinically relevant fatigue, defined as a score of ≥ 4 on the Brief Fatigue Inventory (BFI)
* Have inactive disease, defined as SELENA SLEDAI ≤ 4 AND/OR no hospitalization or addition or increase in dose of corticosteroids, immunosuppressive agents, or antimalarial medications in the last 30 days.
* Have no commonly recognized medical explanations for fatigue (a history of cancer in the previous 5 years -except certain low risk cancer, unstable thyroid disease, moderate to severe chronic kidney disease, moderate to severe anemia)
* Are taking stable doses of anti-malarial therapy (hydroxychloroquine, quinacrine) for at least 6 months.
* Baseline glucocorticoid dose equivalent of ≤ 10 mg prednisone.
* No other planned intervention for fatigue other than current stable medication regimen

Exclusion Criteria:

* Pregnant or breast feeding
* Have a diagnosis of untreated mood disorder, e.g., bipolar or major depressive disorder
* Have an initiation, a cessation or change of treatment of any chronic medications, dietary supplements, behavioral therapy, physical therapy etc., or any planned change of medications, supplements or therapies during the study
* Acupuncture or acupressure receipt in past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women aged 18 years and older
Enrollment: 52 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan
Locations (1):
- Domino's Farms, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zick SM, Sen A, Wyatt GK, Murphy SL, Arnedt JT, Harris RE. Investigation of 2 Types of Self-administered Acupressure for Persistent Cancer-Related Fatigue in Breast Cancer Survivors: A Randomized Clinical Trial. JAMA Oncol. 2016 Nov 1;2(11):1470-1476. doi: 10.1001/jamaoncol.2016.1867. PMID 27388752
- [Background] Zick SM, Wyatt GK, Murphy SL, Arnedt JT, Sen A, Harris RE. Acupressure for persistent cancer-related fatigue in breast cancer survivors (AcuCrft): a study protocol for a randomized controlled trial. BMC Complement Altern Med. 2012 Aug 21;12:132. doi: 10.1186/1472-6882-12-132. PMID 22909076
- [Background] Zick SM, Alrawi S, Merel G, Burris B, Sen A, Litzinger A, Harris RE. Relaxation acupressure reduces persistent cancer-related fatigue. Evid Based Complement Alternat Med. 2011;2011:142913. doi: 10.1155/2011/142913. Epub 2010 Sep 2. PMID 20924499
- [Background] Harris RE, Jeter J, Chan P, Higgins P, Kong FM, Fazel R, Bramson C, Gillespie B. Using acupressure to modify alertness in the classroom: a single-blinded, randomized, cross-over trial. J Altern Complement Med. 2005 Aug;11(4):673-9. doi: 10.1089/acm.2005.11.673. PMID 16131291
- [Background] Danchenko N, Satia JA, Anthony MS. Epidemiology of systemic lupus erythematosus: a comparison of worldwide disease burden. Lupus. 2006;15(5):308-18. doi: 10.1191/0961203306lu2305xx. PMID 16761508
- [Background] Bertsias GK, Salmon JE, Boumpas DT. Therapeutic opportunities in systemic lupus erythematosus: state of the art and prospects for the new decade. Ann Rheum Dis. 2010 Sep;69(9):1603-11. doi: 10.1136/ard.2010.135186. PMID 20699243
- [Background] Cheuk DK, Yeung WF, Chung KF, Wong V. Acupuncture for insomnia. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD005472. doi: 10.1002/14651858.CD005472.pub3. PMID 22972087
- [Background] Frost H, Stewart-Brown S. Acupressure for low back pain. BMJ. 2006 Mar 25;332(7543):680-1. doi: 10.1136/bmj.332.7543.680. No abstract available. PMID 16565098
- [Background] Kim YC, Lee MS, Park E-S, Lew J-H, Lee B-J. Acupressure for the Treatment of Musculoskeletal Pain Conditions: A Systematic Review. Journal of Musculoskeletal Pain 20 (2): 116-121, 2012.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant who was consented but did not actually begin the intervention.
Period: Overall Study
Arm/Group | Relaxing Acupressure Plus Usual Care | Stimulating Acupressure Plus Usual Care | Sham Acupressure Plus Usual Care | Usual Care
Started | 11 | 14 | 14 | 13
Completed | 6 | 3 | 7 | 7
Not Completed | 5 | 11 | 7 | 6
Not completed — Withdrawal by Subject | 5 | 11 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relaxing Acupressure Plus Usual Care | Stimulating Acupressure Plus Usual Care | Sham Acupressure Plus Usual Care | Usual Care | Total
Number analyzed (Participants) | 11 | 14 | 14 | 13 | 52
Age, Continuous [Mean (Full Range); unit: years] | 49.4 [30 to 67] | 47.3 [28 to 74] | 53.3 [40 to 66] | 46.5 [35 to 60] | 49.1 [28 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 14 | 13 | 52
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 14 | 12 | 13 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0
  Black | 2 | 5 | 3 | 4 | 14
  White | 9 | 8 | 10 | 9 | 36
  Asian | 0 | 0 | 0 | 0 | 0
  Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 0 | 1 | 1 | 0 | 2
  Unknown & Refused | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 14 | 14 | 13 | 52
Lupus flare severity categorization [Count of Participants; unit: Participants] — Four categories are: none, mild, moderate, and severe.
  Participants
    No | 5 | 5 | 3 | 4 | 17
    Mild | 2 | 3 | 6 | 3 | 14
    Moderate | 2 | 5 | 4 | 4 | 15
    Severe | 2 | 1 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Severity and Interference
Description: Fatigue severity and interference will be determined according the Brief Fatigue Inventory questionnaire. The Brief Fatigue Inventory (BFI) survey questionnaire is a 9-question survey, with each question having 11 possible answers ("No fatigue" to "As bad as you can imagine"), scored from 0 to 10, with the total score being the sum of a participant's individual questions scores at a timepoint and will range from 0 to 90. Lower scores are considered good, better, or healthy, and increasingly higher scores indicate greater fatigue.
Time Frame: Four weeks post-treatment
Population: This is an intent to treat analysis.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Relaxing Acupressure Plus Usual Care | Stimulating Acupressure Plus Usual Care | Sham Acupressure Plus Usual Care | Usual Care
Number analyzed (Participants) | 11 | 14 | 14 | 13
score on a scale | 3.8 [0.1 to 6.9] | 4.3 [3.4 to 5] | 3.7 [1.4 to 6.8] | 4.6 [2 to 7.9]

2. Secondary Outcome: Quality of Life Satisfaction
Description: Quality of Life will be determined by the Rand SF-36. It is a reliable and valid self-report questionnaire consisting of 36 items aggregated to score 8 subscales related to physical and mental health. Subscales include Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Function, Role Emotional and Mental Health. Each subscale is calibrated to a scale from 0 to 100 where 0 represents worst outcome and 100 represents best possible outcome.
Time Frame: Four weeks post-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Relaxing Acupressure Plus Usual Care | Stimulating Acupressure Plus Usual Care | Sham Acupressure Plus Usual Care | Usual Care
Number analyzed (Participants) | 11 | 14 | 14 | 13
score on a scale
  Physical Functioning | 74.1 [50 to 100] | 53.3 [30 to 80] | 55 [20 to 90] | 66.4 [30 to 100]
  Role Limitations due to physical health | 25 [0 to 100] | 8.3 [0 to 25] | 28.6 [0 to 100] | 39.3 [0 to 100]
  Role limitations due to emotional problems | 38.9 [0 to 100] | 77.8 [33 to 100] | 52.4 [0 to 100] | 80.9 [0 to 100]
  Energy/Fatigue | 38.3 [30 to 55] | 26.7 [20 to 35] | 35.7 [0 to 60] | 31.4 [0 to 80]
  Emotional Well-being | 66 [52 to 88] | 88 [84 to 92] | 76 [56 to 92] | 72.6 [52 to 88]
  Social Functioning | 43.7 [25 to 50] | 54.2 [50 to 62.5] | 55.3 [50 to 75] | 66.1 [50 to 100]
  Pain | 60.4 [32.5 to 90] | 51.6 [32.5 to 67.5] | 65 [22.5 to 100] | 68.2 [32.5 to 100]
  General health | 42.5 [20 to 60] | 43.3 [25 to 75] | 40.7 [20 to 80] | 44.3 [15 to 90]

3. Secondary Outcome: Sleep Quality
Description: Sleep quality will be determined by the Pittsburgh Sleep Quality Index. The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Total scores range from 0 to 21. Higher scores indicate worse sleep quality.
Time Frame: Four weeks post-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Relaxing Acupressure Plus Usual Care | Stimulating Acupressure Plus Usual Care | Sham Acupressure Plus Usual Care | Usual Care
Number analyzed (Participants) | 11 | 14 | 14 | 13
score on a scale | 9.3 [6 to 12] | 9.3 [5 to 12] | 7.6 [4 to 10] | 10.3 [8 to 14]

4. Secondary Outcome: Presence of Pain, Intensity, and Interference
Description: Pain presence, intensity and interference will be determined by the Brief Pain Inventory. The Brief Pain Inventory is an instrument that separately measures pain intensity and interference with physical and emotional functioning, such as sleep, relations with others, and enjoyment of life. Pain intensity is measured on a scale of 0 to 10 where 0 means no pain and 10 means unbearable pain. Pain interference is measured on a scale of 0 - 10, where 0 = does not interfere, 10 = completely interferes.
Time Frame: Four weeks post-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Relaxing Acupressure Plus Usual Care | Stimulating Acupressure Plus Usual Care | Sham Acupressure Plus Usual Care | Usual Care
Number analyzed (Participants) | 11 | 14 | 14 | 13
score on a scale
  Pain intensity | 3.7 [1 to 6.7] | 5 [4.75 to 5.5] | 3.7 [2.5 to 6] | 3.5 [1.25 to 6]
  Pain Interference | 3.09 [0 to 7.4] | 3.8 [2.3 to 4.7] | 3.1 [0.7 to 6.7] | 2.06 [0 to 6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over total of 10 weeks which includes 6 weeks of treatment period and 4 weeks of post-treatment follow-up period.
Arm/Group | Relaxing Acupressure Plus Usual Care | Stimulating Acupressure Plus Usual Care | Sham Acupressure Plus Usual Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 3/11 | 3/14 | 2/14 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relaxing Acupressure Plus Usual Care (N=11) | Stimulating Acupressure Plus Usual Care (N=14) | Sham Acupressure Plus Usual Care (N=14) | Usual Care (N=13)
hospitalized for Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild concussion, hospitalized (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Fall in the bathroom. partially torn ligament.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relaxing Acupressure Plus Usual Care (N=11) | Stimulating Acupressure Plus Usual Care (N=14) | Sham Acupressure Plus Usual Care (N=14) | Usual Care (N=13)
Severe cold and flu (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
outpatient surgery for vericose veins (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pain at accupressure points+minor bruising at points (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sinus cold (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accupressure causing pain in joints of the fingers when applying pressure (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lupus flare (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Nausea, Vomitting and belly pain
Root canal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Dental surgery
Foot surgery for plantar fascitis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lupus flare (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Swelling in knee
Lupus flare up (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — swollen hands, blotches, joint pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT03200548/Prot_SAP_000.pdf